CLINICAL TRIAL: NCT01369576
Title: A Double-blind, Randomized, Parallel Group Study to Determine the Effect of Initial Prescription of Zopiclone on the Level of Compliance With CPAP in Adult Patients Treated for OSA at 26 Weeks
Brief Title: Effect of Zopiclone on Compliance With Continuous Positive Airway Pressure in Obstructive Sleep Apnea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OSR Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OSRM-0511
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — zopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Usual sleep apnea and CPAP care Sleep apnea OSR Medical Treatment Plan©
  Interventions: Drug: Placebo
- zopiclone (Experimental): Sleep apnea OSR Medical Treatment plan ©
  Interventions: Drug: Zopiclone

INTERVENTIONS:
Drug: Placebo — 3.75-7.5mg 14 doses 4 weeks
  Arms: Placebo
Drug: Zopiclone — 3.75-7.5mg 14 doses 4 weeks
  Arms: zopiclone

SUMMARY:
The clinical population targeted will be newly diagnosed patients with polysomnographically diagnosed OSA who are not currently taking hypnotics for concomitantly diagnosed insomnia. Outpatients who are also judged to be capable to follow the study procedures (consent, timelines, visits, questionnaires) and who do not have any concurrent disease that in the view of the investigator will interfere with participation in the trial to completion will be included. Approximately 160 subjects were recruited (80 per treatment arm) in the recent trial of eszopiclone. This size is expected to be able to discern an important difference of 80 minutes per night. In the current clinical population newly prescribed CPAP at Mount Sinai Hospital, the average compliance after 4 weeks of initiation of nCPAP was 4:01 (SD 2:59) hours per night. To be able to discern a difference of at least 1 hour (60 minutes) in usage per night, including entirely non-adherent patients who do not use treatment at all as 'zero hour' users, would require randomization of 264 patients (132 per group).

Our hypothesis for this study is that initial titration of CPAP treatment of OSA may be improved by initial prescription of a common hypnotic, zopiclone. To answer this question we intend to recruit 264 consecutive consenting subjects with OSA confirmed by a physician (ABSM or by a respirologist with extensive sleep medicine experience) with supportive polysomnography results who are willing to initiate long-term CPAP treatment.

DETAILED DESCRIPTION:
Background: Obstructive sleep apnea (OSA) is a common sleep breathing disorder that is associated with serious complications. Continuous positive airway pressure (CPAP) is the treatment of choice for most patients but its use in the real world is limited by low patient adherence which may result in sub-optimal outcomes for some patients. A single hypnotic with low risk of adverse effects is a cost-effective intervention to augment the currently low adherence to CPAP, especially if only prescribed for a limited time. The hypnotic is generic zopiclone 3.75-7.5 mg at bedtime for up to 14 doses.

The clinical population targeted will be newly expert physician-diagnosed patients polysomnographically supported OSA who are not currently taking hypnotics for concomitantly diagnosed insomnia. Outpatients who are also judged to be capable to follow the study procedures (consent, timelines, visits, questionnaires) and who do not have any concurrent disease that in the view of the investigator will interfere with participation in the trial to completion will be included.

ELIGIBILITY:
Inclusion Criteria:

* MD diagnosis of obstructive sleep apnea
* No previous use of CPAP
* No concurrent use of hypnotic medication

Exclusion Criteria:

* Fatal comorbidities (i.e., life expectancy less than 6 months)
* Contraindications for CPAP use
* Pregnancy
* Liver Failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
CPAP adherence | 6 months

SECONDARY OUTCOMES:
ESS and SAQLI scores, changes from baseline, % time of average CPAP usage over the last month/ self-estimated total sleep time (h). Residual AHI monitored, analysed for similar findings at trial closure and analysis, but is not an efficacy parameter | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Verschelden, MD DABSM, Principal Investigator — Cite de la Sante, University of Montreal, OSR Medical, Institut de medecine specialisee de Laval (IMSL); Marcel Baltzan, MDCM DABSM, Principal Investigator — McGill University, OSR Medical, Institut de medecine du sommeil (IMS); Kateri Champagne, MD DABSM, Principal Investigator — McGill University Health Centre (MUHC), OSR Medical, Institut de medecine du sommeil (IMS); Germaine Tanzimat, RN, Principal Investigator — OSR Medical Inc.; Barbara Capozzolo, MSc, Principal Investigator — OSR Medical Inc.
Locations (4):
- Canada (4):
  - Cite de la Sante, Laval, Quebec
  - Institut de medecine specialisee de Laval, Laval, Quebec
  - Institut de Medecine du sommeil, Montreal, Quebec
  - Mount Sinai Hospital, Montreal, Quebec

REFERENCES:
- [Background] Wolkove N, Baltzan M, Kamel H, Dabrusin R, Palayew M. Long-term compliance with continuous positive airway pressure in patients with obstructive sleep apnea. Can Respir J. 2008 Oct;15(7):365-9. doi: 10.1155/2008/534372. PMID 18949106
- [Background] Weaver TE, Grunstein RR. Adherence to continuous positive airway pressure therapy: the challenge to effective treatment. Proc Am Thorac Soc. 2008 Feb 15;5(2):173-8. doi: 10.1513/pats.200708-119MG. PMID 18250209
- [Background] Smith I, Nadig V, Lasserson TJ. Educational, supportive and behavioural interventions to improve usage of continuous positive airway pressure machines for adults with obstructive sleep apnoea. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007736. doi: 10.1002/14651858.CD007736. PMID 19370691
- [Background] Lettieri CJ, Shah AA, Holley AB, Kelly WF, Chang AS, Roop SA; CPAP Promotion and Prognosis-The Army Sleep Apnea Program Trial. Effects of a short course of eszopiclone on continuous positive airway pressure adherence: a randomized trial. Ann Intern Med. 2009 Nov 17;151(10):696-702. doi: 10.7326/0003-4819-151-10-200911170-00006. PMID 19920270
- [Background] Lettieri CJ, Collen JF, Eliasson AH, Quast TM. Sedative use during continuous positive airway pressure titration improves subsequent compliance: a randomized, double-blind, placebo-controlled trial. Chest. 2009 Nov;136(5):1263-1268. doi: 10.1378/chest.09-0811. Epub 2009 Jun 30. PMID 19567493